CLINICAL TRIAL: NCT01196117
Title: Sleepiness and the Effects of CPAP on Salivary Cortisol and Alpha-Amylase Levels in Patients With Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 481-04
Record Dates: First submitted 2010-09-03; First posted 2010-09-08 (Estimated); Results first posted 2020-04-01 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Sleep Apnea; Sleep Disordered Breathing
Keywords: automatic positive airway pressure (APAP); continuous positive airway pressure (CPAP); Salivary Cortisol; Apnea; Sleep Apnea and/or any Sleep Disordered Breathing
MeSH Terms: conditions — Sleep Apnea Syndromes; Apnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 14 days of Placebo therapy, then CPAP (Placebo Comparator): 14 days of placebo therapy - use of guaifenesin with salivary cortisol measurement and Epworth Sleepiness Score (ESS) documentation
  Interventions: Device: 14 days of placebo therapy
- 14 days of CPAP therapy (Active Comparator): 14 days of continuous positive airway pressure (CPAP) therapy with salivary cortisol measurement and Epworth Sleepiness Score (ESS) documentation
  Interventions: Device: 14 days of CPAP therapy

INTERVENTIONS:
Device: 14 days of placebo therapy — 14 days of placebo therapy - use of guaifenesin with salivary cortisol measurement and Epworth Sleepiness Score (ESS) documentation
  Other Names: placebo arm, non-CPAP arm
  Arms: 14 days of Placebo therapy, then CPAP
Device: 14 days of CPAP therapy — 14 days of continuous positive airway pressure (CPAP) therapy with salivary cortisol measurement and Epworth Sleepiness Score (ESS) documentation
  Other Names: CPAP arm
  Arms: 14 days of CPAP therapy

SUMMARY:
Patients with Obstructive Sleep Apnea Syndrome (OSAS) will evidence higher levels of salivary cortisol and alpha-amylase levels prior to use of placebo and continuous positive airway pressure (CPAP) and will evidence a decrease in these levels after consistent use of continuous positive airway pressure (CPAP) therapy as compared to placebo. Their level of sleepiness will also decrease with the use of CPAP therapy and will correlate with the levels of salivary cortisol and alpha-amylase in relation to their subjective sleepiness scale, Psychomotor Vigilance Test (PVT), and pupillometry.

DETAILED DESCRIPTION:
It has been shown that there is an inconsistent response in serum cortisol levels in patients with Obstructive Sleep Apnea Syndrome (OSAS), but it is undetermined whether a change in hormone level was not seen due to compliance issues in these long-term studies. These investigators will be employing compliance monitoring continuous positive airway pressure (CPAP) machines and also assessing "sleepiness" before and after therapy. Sleepiness is the dependent variable in our study and will be measured subjectively using sleepiness scales and objectively using Psychomotor Vigilance Test (PVT) and an autonomic measure using pupillometry prior, during and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Male and female
* Between ages 18 and 90
* Undergo a Polysomnography (PSG) with evidence of any sleep disordered breathing including snoring, mild/moderate/severe sleep apnea, and/or restless legs

Exclusion Criteria:

* Ages 17 and under
* Pregnant women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2004-11-15; Primary Completion 2011-12-15 (Actual); Study Completion 2011-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hersel Raff, PhD, Study Chair — Medical College of Wisconsin; Sandra L Ettema, MD, PhD, Study Chair — Medical College of Wisconsin; Laura Brusky, MD, Study Chair — Medical College of Wisconsin; B Tucker Woodson, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert West Clinics - Otolaryngology Clinc, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Block AJ, Boysen PG, Wynne JW, Hunt LA. Sleep apnea, hypopnea and oxygen desaturation in normal subjects. A strong male predominance. N Engl J Med. 1979 Mar 8;300(10):513-7. doi: 10.1056/NEJM197903083001001. PMID 216912
- [Background] Bradley TD, Phillipson EA. Pathogenesis and pathophysiology of the obstructive sleep apnea syndrome. Med Clin North Am. 1985 Nov;69(6):1169-85. doi: 10.1016/s0025-7125(16)30981-6. PMID 3934481
- [Background] Sullivan CE, Issa FG. Obstructive sleep apnea. Clin Chest Med. 1985 Dec;6(4):633-50. PMID 3936665
- [Background] Pasquali R, Colella P, Cirignotta F, Mondini S, Gerardi R, Buratti P, Rinaldi Ceroni A, Tartari F, Schiavina M, Melchionda N, et al. Treatment of obese patients with obstructive sleep apnea syndrome (OSAS): effect of weight loss and interference of otorhinolaryngoiatric pathology. Int J Obes. 1990 Mar;14(3):207-17. PMID 2341227
- [Background] Onusko E. Diagnosing secondary hypertension. Am Fam Physician. 2003 Jan 1;67(1):67-74. PMID 12537168
- [Background] Weitzman ED, Czeisler CA, Zimmerman JC, Moore-Ede MC. Biological rhythms in man: relationship of sleep-wake, cortisol, growth hormone, and temperature during temporal isolation. Adv Biochem Psychopharmacol. 1981;28:475-99. No abstract available. PMID 7010946
- [Background] Wittels EH. Obesity and hormonal factors in sleep and sleep apnea. Med Clin North Am. 1985 Nov;69(6):1265-80. doi: 10.1016/s0025-7125(16)30986-5. PMID 3906303
- [Background] Entzian P, Linnemann K, Schlaak M, Zabel P. Obstructive sleep apnea syndrome and circadian rhythms of hormones and cytokines. Am J Respir Crit Care Med. 1996 Mar;153(3):1080-6. doi: 10.1164/ajrccm.153.3.8630548.
- [Background] Bratel T, Wennlund A, Carlstrom K. Pituitary reactivity, androgens and catecholamines in obstructive sleep apnoea. Effects of continuous positive airway pressure treatment (CPAP). Respir Med. 1999 Jan;93(1):1-7. doi: 10.1016/s0954-6111(99)90068-9. PMID 10464840
- [Background] Vgontzas AN, Chrousos GP. Sleep, the hypothalamic-pituitary-adrenal axis, and cytokines: multiple interactions and disturbances in sleep disorders. Endocrinol Metab Clin North Am. 2002 Mar;31(1):15-36. doi: 10.1016/s0889-8529(01)00005-6. PMID 12055986
- [Background] Lanfranco F, Gianotti L, Maccario M. Endocrine and metabolic alterations in obstructive sleep apnea syndrome. J Endocrinol Invest. 2003 Jun;26(6):491-2. doi: 10.1007/BF03345208. No abstract available. PMID 12952359
- [Background] Grunstein RR, Handelsman DJ, Lawrence SJ, Blackwell C, Caterson ID, Sullivan CE. Neuroendocrine dysfunction in sleep apnea: reversal by continuous positive airways pressure therapy. J Clin Endocrinol Metab. 1989 Feb;68(2):352-8. doi: 10.1210/jcem-68-2-352. PMID 2493027
- [Background] Cooper BG, White JE, Ashworth LA, Alberti KG, Gibson GJ. Hormonal and metabolic profiles in subjects with obstructive sleep apnea syndrome and the acute effects of nasal continuous positive airway pressure (CPAP) treatment. Sleep. 1995 Apr;18(3):172-9. PMID 7610313
- [Background] Grunstein RR, Stewart DA, Lloyd H, Akinci M, Cheng N, Sullivan CE. Acute withdrawal of nasal CPAP in obstructive sleep apnea does not cause a rise in stress hormones. Sleep. 1996 Dec;19(10):774-82. doi: 10.1093/sleep/19.10.774. PMID 9085485
- [Background] Meston N, Davies RJ, Mullins R, Jenkinson C, Wass JA, Stradling JR. Endocrine effects of nasal continuous positive airway pressure in male patients with obstructive sleep apnoea. J Intern Med. 2003 Nov;254(5):447-54. doi: 10.1046/j.1365-2796.2003.01212.x. PMID 14535966
- [Background] Greenberg HE, Rapoport DM, Rothenberg SA, Kanengiser LA, Norman RG, Goldring RM. Endogenous opiates modulate the postapnea ventilatory response in the obstructive sleep apnea syndrome. Am Rev Respir Dis. 1991 Jun;143(6):1282-7. doi: 10.1164/ajrccm/143.6.1282. PMID 2048814
- [Background] Follenius M, Krieger J, Krauth MO, Sforza F, Brandenberger G. Obstructive sleep apnea treatment: peripheral and central effects on plasma renin activity and aldosterone. Sleep. 1991 Jun;14(3):211-7. PMID 1896722
- [Background] Raff H: Salivary cortisol: a useful measurement in the diagnosis of cushing's syndrome and the evaluation of the hypothalamic-pituitary-adrenal axis. The Endocrinologist 2000; 10: 9-17
- [Background] Laudat MH, Cerdas S, Fournier C, Guiban D, Guilhaume B, Luton JP. Salivary cortisol measurement: a practical approach to assess pituitary-adrenal function. J Clin Endocrinol Metab. 1988 Feb;66(2):343-8. doi: 10.1210/jcem-66-2-343. PMID 2828410
- [Background] Papanicolaou DA, Mullen N, Kyrou I, Nieman LK. Nighttime salivary cortisol: a useful test for the diagnosis of Cushing's syndrome. J Clin Endocrinol Metab. 2002 Oct;87(10):4515-21. doi: 10.1210/jc.2002-020534. PMID 12364428
- [Background] Raff H, Findling JW. A physiologic approach to diagnosis of the Cushing syndrome. Ann Intern Med. 2003 Jun 17;138(12):980-91. doi: 10.7326/0003-4819-138-12-200306170-00010. No abstract available. PMID 12809455
- [Background] Umeda T, Hiramatsu R, Iwaoka T, Shimada T, Miura F, Sato T. Use of saliva for monitoring unbound free cortisol levels in serum. Clin Chim Acta. 1981 Mar 5;110(2-3):245-53. doi: 10.1016/0009-8981(81)90353-3. PMID 6261989
- [Background] Vining RF, McGinley RA, Maksvytis JJ, Ho KY. Salivary cortisol: a better measure of adrenal cortical function than serum cortisol. Ann Clin Biochem. 1983 Nov;20 (Pt 6):329-35. doi: 10.1177/000456328302000601. PMID 6316831
- [Background] Raff H, Raff JL, Findling JW. Late-night salivary cortisol as a screening test for Cushing's syndrome. J Clin Endocrinol Metab. 1998 Aug;83(8):2681-6. doi: 10.1210/jcem.83.8.4936. PMID 9709931
- [Background] Castro M, Elias PC, Martinelli CE Jr, Antonini SR, Santiago L, Moreira AC. Salivary cortisol as a tool for physiological studies and diagnostic strategies. Braz J Med Biol Res. 2000 Oct;33(10):1171-5. doi: 10.1590/s0100-879x2000001000006. PMID 11004717
- [Background] Broderick JE, Arnold D, Kudielka BM, Kirschbaum C. Salivary cortisol sampling compliance: comparison of patients and healthy volunteers. Psychoneuroendocrinology. 2004 Jun;29(5):636-50. doi: 10.1016/S0306-4530(03)00093-3. PMID 15041086
- [Background] Chatterton RT Jr, Vogelsong KM, Lu YC, Ellman AB, Hudgens GA. Salivary alpha-amylase as a measure of endogenous adrenergic activity. Clin Physiol. 1996 Jul;16(4):433-48. doi: 10.1111/j.1475-097x.1996.tb00731.x. PMID 8842578
- [Background] Skosnik PD, Chatterton RT Jr, Swisher T, Park S. Modulation of attentional inhibition by norepinephrine and cortisol after psychological stress. Int J Psychophysiol. 2000 Apr;36(1):59-68. doi: 10.1016/s0167-8760(99)00100-2. PMID 10700623
- [Background] Nater UM, Rohleder N, Gaab J, Berger S, Jud A, Kirschbaum C, Ehlert U. Human salivary alpha-amylase reactivity in a psychosocial stress paradigm. Int J Psychophysiol. 2005 Mar;55(3):333-42. doi: 10.1016/j.ijpsycho.2004.09.009. PMID 15708646
- [Background] Nater UM, La Marca R, Florin L, Koller MM, Ehlert U: The relationship between salivary alpha-amylase and plasma catecholamines. J Psychophysiol 2003; 17(3): 170 (abstract).
- [Background] Graeber RC: Aircrew fatigue and circadian rhythmicity. In: Wiener E, Nagel DC, eds. Human Factors in Aviation. New York: Academic Press; 1987: 1-48
- [Background] Akerstedt T. Sleepiness as a consequence of shift work. Sleep. 1988 Feb;11(1):17-34. doi: 10.1093/sleep/11.1.17. PMID 3283910
- [Background] Price WJ, Holley DC. Shiftwork and safety in aviation. Occup Med. 1990 Apr-Jun;5(2):343-77. PMID 2203162
- [Background] Kecklund G, Akerstedt T. Sleepiness in long distance truck driving: an ambulatory EEG study of night driving. Ergonomics. 1993 Sep;36(9):1007-17. doi: 10.1080/00140139308967973. PMID 8404830
- [Background] Akerstedt T. Work hours and sleepiness. Neurophysiol Clin. 1995;25(6):367-75. doi: 10.1016/0987-7053(96)84910-0. PMID 8904199
- [Background] Mitler MM, Miller JC, Lipsitz JJ, Walsh JK, Wylie CD. The sleep of long-haul truck drivers. N Engl J Med. 1997 Sep 11;337(11):755-61. doi: 10.1056/NEJM199709113371106. PMID 9287232
- [Background] Ohayon MM, Caulet M, Philip P, Guilleminault C, Priest RG. How sleep and mental disorders are related to complaints of daytime sleepiness. Arch Intern Med. 1997 Dec 8-22;157(22):2645-52. PMID 9531234
- [Background] Hoddes E, Zarcone V, Smythe H, Phillips R, Dement WC. Quantification of sleepiness: a new approach. Psychophysiology. 1973 Jul;10(4):431-6. doi: 10.1111/j.1469-8986.1973.tb00801.x. No abstract available. PMID 4719486
- [Background] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888
- [Background] Chervin RD, Aldrich MS, Pickett R, Guilleminault C. Comparison of the results of the Epworth Sleepiness Scale and the Multiple Sleep Latency Test. J Psychosom Res. 1997 Feb;42(2):145-55. doi: 10.1016/s0022-3999(96)00239-5. PMID 9076642
- [Background] Jokinen T, Salmi T, Ylikoski A, Partinen M. Use of computerized visual performance test in assessing day-time vigilance in patients with sleep apneas and restless sleep. Int J Clin Monit Comput. 1995;12(4):225-30. doi: 10.1007/BF01207203. PMID 8820329
- [Background] Loh S, Lamond N, Dorrian J, Roach G, Dawson D. The validity of psychomotor vigilance tasks of less than 10-minute duration. Behav Res Methods Instrum Comput. 2004 May;36(2):339-46. doi: 10.3758/bf03195580. PMID 15354700
- [Background] Lowenstein O, Feinberg R, Loewenfeld ID: Pupillary movements during acute and chronic fatigue. Investigative Ophthalmolog 1963; 2: 138-157
- [Background] Yoss RE, Moyer NJ, Ogle KN. The pupillogram and narcolepsy. A method to measure decreased levels of wakefulness. Neurology. 1969 Oct;19(10):921-8. doi: 10.1212/wnl.19.10.921. No abstract available. PMID 5387594
- [Background] Ludtke H, Wilhelm B, Adler M, Schaeffel F, Wilhelm H. Mathematical procedures in data recording and processing of pupillary fatigue waves. Vision Res. 1998 Oct;38(19):2889-96. doi: 10.1016/s0042-6989(98)00081-9. PMID 9797985
- [Background] Merrit SL, Schnyders HC, Mercer P: Circadian aspects of papillary unrest reflecting daytime sleepiness. Sleep Research Online 1999; 2(Sup 1): 773
- [Background] Merrit SL, Schnyders HC, Mercer P, Zhou X: The sensitivity of pupillography to circadian aspects of sleepiness. J Sleep Research 1998; 7(Sup 2): 176
- [Derived] Raff H, Ettema SL, Eastwood DC, Woodson BT. Salivary cortisol in obstructive sleep apnea: the effect of CPAP. Endocrine. 2011 Aug;40(1):137-9. doi: 10.1007/s12020-011-9474-1. Epub 2011 Apr 26. No abstract available. PMID 21519909

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from sleep clinic patients scheduled for polysomnography.
Pre-assignment Details: Participants without prior treatment of obstructive sleep apnea (OSA) or overt airway structural pathology that would interfere with continuous positive airway pressure (CPAP) were recruited.
Groups:
- 14 Days of Continuous Positive Airway Pressure (CPAP) Therapy: 14 days of continuous positive airway pressure (CPAP) therapy with salivary cortisol measurement and Epworth Sleepiness Score (ESS) documentation
Period: Placebo, Then CPAP
Arm/Group | 14 Days of Placebo Therapy | 14 Days of Continuous Positive Airway Pressure (CPAP) Therapy
Started | 18 | 0
Completed | 18 | 0
Not Completed | 0 | 0
Period: CPAP
Arm/Group | 14 Days of Placebo Therapy | 14 Days of Continuous Positive Airway Pressure (CPAP) Therapy
Started | 0 | 18
Completed | 0 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants received 14 days of placebo therapy then 14 days of continuous positive airway pressure (CPAP) therapy
Arm/Group | All Study Participants
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 9
Apnea-hyponea Index (AHI) [Mean (Standard Deviation); unit: units on a scale] — AHI<5 Normal <=5 AHI <15 Mild Sleep Apnea 15<= AHI <30 Moderate Sleep Apnea AHI>=30 Severe Sleep Apnea
  units on a scale | 30.8 (32.1)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — <18.5 Underweight range >=18.5 BMI <24.9 Healthy weight range >25.0 BMI < 29.9 Overweight range >30.0 BMI <29.9 Obese weight range
  kg/m^2 | 33.8 (6.2)

OUTCOME MEASURES:

1. Primary Outcome: Salivary Cortisol Level
Description: Salivary Cortisol was measured by enzyme-linked immunosorbent assay. The reference range for healthy adults is <4.2 nmol/l. Samples were collected at ~7am and ~11pm on each Day: 0, 1, 7 and 14 through a salivary swab.
Time Frame: Difference between Baseline(Day 0) and Average of Day 1,7,14.
Population: We have made a best faith effort from a manuscript to determine the primary outcome measure; Salivary Cortisol Level; but access to the primary data has been lost and it additionally cannot be found in the manuscript. Despite all efforts to contact the PI/study team members, the statisticians and date are gone.
Groups:
- 14 Days of CPAP Therapy: 14 days of continuous positive airway pressure (CPAP) therapy with salivary cortisol measurement
Arm/Group | 14 Days of Placebo Therapy | 14 Days of CPAP Therapy
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Epworth Sleepiness Score (ESS)
Description: Epworth Sleepiness Score (ESS) is a scale to assess sleepiness during waking hours. The scale ranges from 0-24 with higher scores indicative of greater sleepiness.
Time Frame: Difference between Baseline(Day 0) and Average of Day 1,7,14.
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | 14 Days of Placebo Therapy, Then CPAP | 14 Days of CPAP Therapy
Number analyzed (Participants) | 18 | 18
units on a scale | 10.7 [8.5 to 12.9] | 8.9 [6.8 to 11.2]
Statistical Analysis 1: Comparison: 14 Days of Placebo Therapy, Then CPAP vs 14 Days of CPAP Therapy; Test type: Superiority; p = 0.0009, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Salivary Cortisol in Participants Who Used Continuous Positive Airway Pressure (CPAP) at ~7am, Day 0
Description: Salivary Cortisol was measured by enzyme-linked immunosorbent assay. The reference range for healthy adults is <4.2 nmol/l.
Time Frame: Day 0, 7am
Population: A sub-analysis was performed on those using CPAP>= 3 hours per night compared to those who used CPAP< 3 hours per night
Measure: Median (95% Confidence Interval); unit: nmol/l
Groups:
- CPAP>= 3 Hours Per Night: The average nightly CPAP use in the group using CPAP for >=3 hours (N=9) was 311 minutes (180-444) minutes.
- CPAP<3 Hours Per Night: In the group using CPAP for <3hours (N=9), it was 33 minutes (2-85) minutes.
Arm/Group | CPAP>= 3 Hours Per Night | CPAP<3 Hours Per Night
Number analyzed (Participants) | 9 | 9
nmol/l | 12.5 [7.6 to 20.8] | 12.1 [7.2 to 20.5]
Statistical Analysis 1: Comparison: CPAP>= 3 Hours Per Night vs CPAP<3 Hours Per Night; Test type: Superiority; p = 0.8938, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Salivary Cortisol in Participants Who Used Continuous Positive Airway Pressure (CPAP) at ~11pm, Day 0
Description: as for outcome 3
Time Frame: Day 0, 11pm
Population: A sub-analysis was performed on those using CPAP>= 3 hours per night compared to those who used CPAP< 3 hours per night
Measure: Median (95% Confidence Interval); unit: nmol/l
Arm/Group | CPAP>= 3 Hours Per Night | CPAP<3 Hours Per Night
Number analyzed (Participants) | 9 | 9
nmol/l | 3.2 [1.6 to 6.4] | 1.2 [0.6 to 2.6]
Statistical Analysis 1: Comparison: CPAP>= 3 Hours Per Night vs CPAP<3 Hours Per Night; Test type: Superiority; p < 0.014, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Salivary Cortisol in Participants Who Used Continuous Positive Airway Pressure (CPAP) at ~7am, Day 1
Description: as for outcome 3
Time Frame: Day 1, 7am
Population: A sub-analysis was performed on those using CPAP>= 3 hours per night compared to those who used CPAP< 3 hours per night
Measure: Median (95% Confidence Interval); unit: nmol/l
Arm/Group | CPAP>= 3 Hours Per Night | CPAP<3 Hours Per Night
Number analyzed (Participants) | 9 | 9
nmol/l | 7.4 [4.4 to 12.2] | 13.6 [8.1 to 23.0]
Statistical Analysis 1: Comparison: CPAP>= 3 Hours Per Night vs CPAP<3 Hours Per Night; Test type: Superiority; p < 0.0200, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Salivary Cortisol in Participants Who Used Continuous Positive Airway Pressure (CPAP) at ~11pm, Day 1
Description: as for outcome 3
Time Frame: Day 1, 11pm
Population: A sub-analysis was performed on those using CPAP>= 3 hours per night compared to those who used CPAP< 3 hours per night
Measure: Median (95% Confidence Interval); unit: nmol/l
Arm/Group | CPAP>= 3 Hours Per Night | CPAP<3 Hours Per Night
Number analyzed (Participants) | 9 | 9
nmol/l | 2.2 [1.1 to 4.4] | 1.8 [0.9 to 3.7]
Statistical Analysis 1: Comparison: CPAP>= 3 Hours Per Night vs CPAP<3 Hours Per Night; Test type: Superiority; p = 0.1321, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Salivary Cortisol in Participants Who Used Continuous Positive Airway Pressure (CPAP) at ~ 7am, Day 7
Description: as for outcome 3
Time Frame: Day 7, 7am
Population: A sub-analysis was performed on those using CPAP>= 3 hours per night compared to those who used CPAP< 3 hours per night
Measure: Mean (95% Confidence Interval); unit: nmol/l
Arm/Group | CPAP>= 3 Hours Per Night | CPAP<3 Hours Per Night
Number analyzed (Participants) | 9 | 9
nmol/l | 9.9 [6.0 to 16.4] | 13.3 [7.9 to 22.3]
Statistical Analysis 1: Comparison: CPAP>= 3 Hours Per Night vs CPAP<3 Hours Per Night; Test type: Superiority; p < 0.2490, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Salivary Cortisol in Participants Who Used Continuous Positive Airway Pressure (CPAP) at ~11pm, Day 7
Description: as for outcome 3
Time Frame: Day 7, 11pm
Measure: Median (95% Confidence Interval); unit: nmol/l
Arm/Group | CPAP>= 3 Hours Per Night | CPAP<3 Hours Per Night
Number analyzed (Participants) | 9 | 9
nmol/l | 3.0 [1.5 to 6.1] | 2.5 [1.2 to 5.1]
Statistical Analysis 1: Comparison: CPAP>= 3 Hours Per Night vs CPAP<3 Hours Per Night; Test type: Superiority; p = 0.5139, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Salivary Cortisol in Participants Who Used Continuous Positive Airway Pressure (CPAP) at ~7am, Day 14
Description: as for outcome 3
Time Frame: Day 14, 7am
Population: A sub-analysis was performed on those using CPAP>= 3 hours per night compared to those who used CPAP< 3 hours per night
Measure: Median (95% Confidence Interval); unit: nmol/l
Arm/Group | CPAP>= 3 Hours Per Night | CPAP<3 Hours Per Night
Number analyzed (Participants) | 9 | 9
nmol/l | 9.2 [5.6 to 15.3] | 15.0 [8.9 to 25.3]
Statistical Analysis 1: Comparison: CPAP>= 3 Hours Per Night vs CPAP<3 Hours Per Night; Test type: Superiority; p = 0.0597, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Salivary Cortisol in Participants Who Used Continuous Positive Airway Pressure (CPAP) at ~11pm, Day 14
Description: as for outcome 3
Time Frame: Day 14, 11pm
Population: A sub-analysis was performed on those using CPAP>= 3 hours per night compared to those who used CPAP< 3 hours per night
Measure: Median (95% Confidence Interval); unit: nmol/l
Arm/Group | CPAP>= 3 Hours Per Night | CPAP<3 Hours Per Night
Number analyzed (Participants) | 9 | 9
nmol/l | 1.9 [1.0 to 4.0] | 2.2 [1.0 to 4.5]
Statistical Analysis 1: Comparison: CPAP>= 3 Hours Per Night vs CPAP<3 Hours Per Night; Test type: Superiority; p = 0.2134, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse Events were observed in a non-systematic way over the course of approximately 6 years the patients were enrolled.
Description: Given the minimal risk nature of this study, adverse events were collected via a non-systematic assessment. The primary risks were loss of confidentiality, some possible discomfort from the mask and the possibility of an adverse event related to the mucolytic, guaifenesin. None of these possible adverse events occurred and they were not collected in a systematic way.
Groups:
- 14 Days of Placebo Therapy, Then CPAP: 14 days of placebo therapy: 14 days of placebo therapy then 14 days of continuous positive airway pressure (CPAP) therapy
- 14 Days of CPAP Therapy: 14 days of continuous positive airway pressure (CPAP) therapy
Arm/Group | 14 Days of Placebo Therapy, Then CPAP | 14 Days of CPAP Therapy
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

LIMITATIONS AND CAVEATS:
The limitation of this trial is the results were entered strictly from a manuscript published in 2011. Despite repeated attempts to reach out, the original study team members, statisticians and data are no longer available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No